CLINICAL TRIAL: NCT05977595
Title: A Descriptive Study of the Cosmetic and Functional Sequelae of Patients Who Received Releasing Incisions in the Management of Acute Upper Limb Burns.
Brief Title: Cosmetic and Functional Sequelae in Hand Burns.
Acronym: AdipoSCAR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL23_0747
Record Dates: First submitted 2023-07-26; First posted 2023-08-04 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-07

CONDITIONS: Hand Burn
Keywords: burns; hands; functional outcomes; skin graft; releasing incisions
MeSH Terms: conditions — Burns

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Deep hand burns: Adult subjects, who were hospitalized at the Pierre Colson Burn Center with a hand burn that required releasing incisions.
  Interventions: Other: Quick DASH Score Visual Analog Scale Scar quality Healing Number of surgeries

INTERVENTIONS:
Other: Quick DASH Score Visual Analog Scale Scar quality Healing Number of surgeries — Functional and aesthetic criteria : Quick DASH Score at 3 month and 6 months, Visual Analog Scale at 3 month and 6 months, scar quality (assessment by surgeon), healing (discontinuation of dressings), need for a second surgical procedure.

SUMMARY:
Although it represents a small percentage of the body surface, the hand is the most exposed part of the body after the face and neck and is one of the area's most frequently involved in burns. It has a social function, but above all, a functionnal one. An optimized reconstruction of this area after the burn allow the patient to recover the best possible function and increase his chances of returning to professional activity and daily life. Advances in burn treatment, such as improved resuscitation management, rapid excision of burns, skin grafting, regular dressings, and improved metabolic support, have reduced the morbidity and mortality of severe burns. However, significant challenges remain.

The hand is the most frequently involved area in burns and is affected in 90% of severe burns. Hand burns requiring releasing incisions are circular, deep burns and represent a significant functional challenge. In the acute setting, current treatment options must prevent complications associated with disruption of the skin's protective function. In the longer term, these treatments should allow the regeneration of fully functional skin. However, some sequelae may persist in the form of sensory deficits, residual pain, retractile scars hindering function in this highly mobile area, or even aesthetic sequelae.

The aim of our study was to perform a descriptive analysis of the aesthetic and functional sequelae related to hand burns that required acute realeasing incisions using objective and subjective tools available in the medical records (demographic, clinical and follow-up data in the context of routine care). This retrospective, non-interventional, data-driven study would provide an overview of the sequelae of hand burns with current therapies.

ELIGIBILITY:
* Inclusion Criteria :

  * Adult patients
  * Acute burn (less than 3 days)
  * Burns of one or both hands or finger burns
  * Skin surface burned less than 40% of the body
  * Chemical, thermal, or electrical burns of the hand.
  * Burn that required a skin graft.
* Exclusion Criteria :

  * Patient refusal
  * Less than 1 month follow-up or death within the first month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult subjects, who were hospitalized at the Pierre Colson Burn Center (University Hospital) with a hand burn that required discharge incisions between January 2019 and June 2023.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Functional score | Through the completion of study, average 6 months
  Functional recovery at 3 months and 6 months after the burn (functional score, return to activities) Healing time (discontinuation of dressings). Scar quality (hypertrophic, retractile, surgical revision necessary and surgery of sequela).
  Burn VAS (1-10) at 3 and 6 months. QuickDASH Score at 3 and 6 months. Scar quality at 6 months. Burn VAS at 3 months and 6 months.
Healing assessment | Through the completion of study, average 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Edouard Herriot University hospital, Lyon, France